CLINICAL TRIAL: NCT07105735
Title: An Exploratory Clinical Study on Allogeneic CAR-T Cell (RN1201) Injection for Autoimmune Diseases Refractory to Standard Therapies
Brief Title: RN1201 Injection for Autoimmune Diseases Refractory to Standard Therapies
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Rui Therapeutics Co., Ltd (Industry); Allorunning Therapeutics (Industry)
Responsible Party: Principal Investigator, Lei Fan, Director of lymphoma center, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RN1201-AID
Record Dates: First submitted 2025-07-24; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Diseases Refractory to Standard Therapies
Keywords: Autoimmune Diseases; Refractory to Standard Therapies
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- allogeneic CAR-T cell therapy (Experimental): RN1201 cells injection will be infused only once intravenously at day 0
  Interventions: Biological: allogeneic CAR-T

INTERVENTIONS:
Biological: allogeneic CAR-T — Fludarabine injection (30 mg/m2，QD×3d) and cyclophosphamide injection (300 mg/m2，QD×3d)will be used to remove the lymphocyte before RN1201 infusion.

SUMMARY:
This is a open-label, exploratory trial to evaluate the safety, feasibility, and preliminary efficacy of RN1201, an Allogeneic CAR-T cell therapy, in patients with autoimmune diseases refractory to standard treatment. Eligible patients with moderate to severe activity of diseases will receive a single infusion of RN1201 following lymphodepletion. Primary endpoints include dose-limiting toxicity and treatment-emergent adverse events. Secondary and exploratory endpoints assess clinical response and cell pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria

1. Voluntary signed informed consent demonstrating understanding of the study and willingness/ability to comply with all trial procedures.
2. Age ≥18 years; both sexes eligible.
3. Documented diagnosis of an autoimmune disease for ≥6 months at screening, including but not limited to immune thrombocytopenia (ITP), autoimmune hemolytic anemia (AIHA), systemic lupus erythematosus (SLE), immune-mediated necrotizing myopathy (IMNM), neuromyelitis optica spectrum disorder (NMOSD), multiple sclerosis (MS), myasthenia gravis (MG), etc.
4. Standard-of-care therapy for ≥8 weeks before screening without achieving complete remission or adequate disease control, with stable dose for >2 weeks.
5. Subjects on corticosteroid monotherapy at screening must be receiving ≥7.5 mg/day prednisone (or equivalent).
6. Disease activity score meeting criteria for moderate-to-severe active disease.
7. Adequate bone-marrow reserve, coagulation, cardiopulmonary, hepatic, and renal function.
8. Agreement to use effective contraception for 24 months after study enrollment.

Exclusion Criteria

Subjects meeting any of the following cannot be enrolled:

1. Known hypersensitivity, allergy, intolerance, or contraindication to RN1201 or any study drug component (fludarabine, cyclophosphamide, tocilizumab) or history of severe allergic reactions.
2. Severe cardiovascular disease or organ failure.
3. Active or uncontrolled infection requiring IV antibiotics or evidence of severe active infection.
4. Significant bleeding tendency (e.g., Gastrointestinal bleeding, coagulopathy, hypersplenism).
5. Hepatitis C virus, HIV, or syphilis infection.
6. History of epilepsy or severe neurological disorders/pathology not attributable to autoimmune disease.
7. Malignancy within 2 years before screening, except adequately treated carcinoma in situ of skin, cervix, or lung or other non-active tumors.
8. Prior CAR-T therapy or other genetically modified T-cell therapy.
9. Prednisone (or equivalent) ≥100 mg/day for ≥14 days within 4 weeks before screening.
10. Pregnancy, lactation, or planned pregnancy within 2 years.
11. Any condition that, in the investigator's judgment, may increase subject risk or interfere with study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of treatment-emergent adverse events (TEAEs) and dose-limiting toxicities (DLTs) | DLTs: Within 28 days after CAR-T cell infusion; TEAEs: From infusion up to 12 months post-treatment.
  TEAEs and DLTs will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) consensus criteria

SECONDARY OUTCOMES:
Objective Response Rate (ORR), Disease control rate (DCR) | Week 4, Month 3, Month 6 and Month 12
  The responses will be assessed by predefined disease specific criteria.
Pharmacokinetic (PK) of RN1201 | up to 12 months
  Levels of CAR-positive T cells in the blood and/or bone marrow
Pharmacodynamic (PD) of RN1201 | up to 12 months
  Levels of B cells and related immune markers (e.g., serum immunoglobulins, autoantibodies) in peripheral blood and/or bone marrow, as indicators of B cell activity and depletion.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Fan, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No